CLINICAL TRIAL: NCT06414590
Title: Neoadjuvant Tebentafusp in Patients With Locally Advanced, Unresectable Primary Uveal Melanoma
Brief Title: Neoadjuvant Tebentafusp for Uveal Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iRISID-2023-2369; JT 33504 (Other: JeffTrial Number)
Record Dates: First submitted 2024-03-25; First posted 2024-05-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Unresectable Uveal Melanoma
Keywords: Neoadjuvant Tebentafusp; Uveal Melanoma; Primary Uveal Melanoma; Neoadjuvant IMCgp100; gp100 peptide-HLA-directed CD3 T cell engager; HLA-A*02:01; KIMMTRAK®; Tebentafusp-tebn; IMCgp100; radioactive plaque therapy; enucleation; radioactive plaque; fine-needle aspiration; circulating tumor-derived DNA; Phase II; advanced primary uveal melanoma; Simon's two stage design
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Tebentafusp in Patients Locally Advanced, Unresectable Primary Uveal Melanoma (Experimental): Tebentafusp administration: 20mcg on Day 1, 30mcg on Day 8, 68 mcg on Day 15, and weekly doses of 68 mcg thereafter. Eye evaluations including clinical examination, ophthalmic ultrasound, optical coherence tomography, and wide-angle fundus imaging will be performed at baseline, Cycle 1 day 1, Cycle 1 day 8, Cycle 2 day 1, prior to definitive treatment for primary uveal melanoma (post-Tebentafusp), and at post-eye treatment evaluation at 3 months. Additionally optical coherence tomography angiography, autofluorescence, fluorescein angiography and MRI orbit will be performed at baseline, post-tebentafusp, and at post-eye treatment evaluation. Blood circulating tumor-derived DNA will be performed at baseline, Cycle 2 day 1, post-Tebentafusp, and at post-eye treatment evaluation at 3 months. Primary eye tumor biopsy (collected by fine-needle aspiration) and aqueous circulating tumor-derived DNA will be performed at baseline and post-Tebentafusp.
  Interventions: Drug: Tebentafusp-Tebn

INTERVENTIONS:
Drug: Tebentafusp-Tebn — Tebentafusp will be administered as follows: 20mcg on Day 1, 30mcg on Day 8, 68 mcg on Day 15, and weekly doses of 68 mcg thereafter.
  Other Names: KIMMTRAK®; IMCgp100; gp100 peptide-HLA-directed CD3 T cell engager

SUMMARY:
This phase II trial tests how well tebentafusp works to shrink tumors prior to primary treatment with surgery or radiation in patients with uveal (eye) melanoma that has spread to nearby tissue or lymph nodes (locally advanced) or that cannot be removed by surgery (unresectable). Tebentafusp is a drug that binds to melanoma tumor cells as well as immune cells called T-cells. This binding causes an immune response against the melanoma cells, which leads to tumor cell death. Tebentafusp has been approved for the treatment of locally advanced and unresectable uveal melanoma. Giving tebentafusp before primary treatment with surgery or radiation may help shrink the tumor, prevent the disease from spreading, or reduce the likelihood that patients will require total eye removal (called enucleation).

DETAILED DESCRIPTION:
This is a prospective, single arm, phase II clinical trial of neoadjuvant Tebentafusp (KIMMTRAK®) in patients with locally advanced primary uveal melanoma. Patients must be HLA-A*02:01 with large, surgically unresectable (other than complete enucleation of the eye) primary uveal melanoma. The efficacy of this treatment will be assessed with the Simon's two stage design. The choice of design is guided by a desire to stop the trial early if the actual regression rate of primary uveal melanoma is 1% or lower.

PRIMARY OBJECTIVE:

I. To assess the efficacy of neoadjuvant tebentafusp in patients with large surgically unresectable (other than complete enucleation of eye) primary uveal melanoma.

SECONDARY OBJECTIVES:

I. To assess the local (eye) and systemic toxicity with tebentafusp treatment. II. To investigate the usefulness of circulating tumor-derived deoxyribonucleic acid (DNA) (ctDNA) as a biomarker for response.

EXPLORATORY OBJECTIVES:

I. To assess sight preservation. II. To assess the change in radiation dose to the fovea.

OUTLINE:

Participants may be screened at Wills Eye Hospital before being consented and treated at Thomas Jefferson University. Patients receive tebentafusp intravenously (IV) over 15-20 minutes on days 1, 8, 15, and 22 of each cycle. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Within 28 days of their last dose of tebentafusp, patients undergo standard of care (SOC) primary eye treatment (plaque radiotherapy or eye enucleation), as decided by their treating physician. Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) at screening, ophthalmic ultrasound, optical coherence tomography (OCT), wide-angle fundus imaging, OCT angiography (OCTA), fluorescein angiography, orbit magnetic resonance imaging (MRI), and collection of blood samples throughout the trial, undergo biopsy and collection of aqueous humour samples at screening and on study, and undergo abdominal MRI and chest and pelvis computed tomography (CT) at screening and during follow up.

After completion of primary eye treatment, patients are followed up at 3 months and then every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient age ≥ 18 years of age at the time of informed consent.
2. Ability to provide and understand written informed consent prior to any study procedures.
3. Willingness to undergo tumor biopsies at baseline and post-Tebentafusp treatment.
4. Treatment naïve primary uveal melanoma with T3 or T4 category tumor size that are surgically unresectable (other than complete enucleation of eye).
5. No surgical indication to completely remove the tumor without enucleation.
6. Clinically or cytologically confirmed primary uveal melanoma.
7. Participants must be HLA-A*02:01 positive.
8. Predicted life expectancy of at least 12 weeks as estimated by investigator
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening.
10. All other relevant medical conditions must be well-managed and stable, in the opinion of the investigator, for at least 28 days prior to first administration of study drug.
11. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

1. Symptomatic uveal melanoma that requires immediate ophthalmological intervention such as enucleation.
2. Evidence of metastatic disease.
3. Previous treatment with Tebentafusp.
4. Patients with any out-of-range laboratory values defined as:

   * Serum creatinine > 1.5 x upper limit of normal (ULN) and/or creatinine clearance (calculated using Cockcroft-Gault Formula, or measured) < 50 mL/minute
   * Albumin < 3.0 g/dl
   * Total bilirubin >1.5 mg/dL (or 1.3 x ULN). Patients with hyperbilirubinemia clinically consistent with an inherited disorder of bilirubin metabolism (e.g., Gilbert syndrome) will be eligible at the discretion of the treating physician and/or the principal investigator.
   * Alanine aminotransferase > 1.5 x ULN
   * Aspartate aminotransferase > 1.5 x ULN
   * Absolute neutrophil count < 1.0 x 109 /L
   * Absolute lymphocyte count < 0.5 x 109 /L
   * Platelet count < 100 x 109 /L
   * Hemoglobin < 9.0 g/dL
   * Uncorrectable abnormal potassium, magnesium, corrected calcium or phosphate abnormality of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0) > grade 1
   * Morning cortisol < lower limit of normal (unless the patient has asymptomatic adrenal insufficiency and is receiving stable replacement doses)
5. History of severe hypersensitivity reactions (eg, anaphylaxis) to other biologic drugs or monoclonal antibodies.
6. Clinically significant cardiac disease or impaired cardiac function, including any of the following:

   * Left Ventricular Ejection Fraction <50%
   * Clinically significant and/or uncontrolled heart disease such as congestive heart failure (New York Heart Association grade ≥ 2), uncontrolled hypertension, or clinically significant arrhythmia uncontrolled with medical treatment
   * QTcF > 470 msec on screening electrocardiogram (ECG) or congenital long QT syndrome
   * Acute myocardial infarction or unstable angina pectoris < 6 months to Screening
7. Active infection requiring systemic antibiotic therapy. Patients requiring systemic antibiotics for infection must have completed therapy at least 1 week prior to the first dose of study drug.
8. Participants with a history of human immunodeficiency virus (HIV) infection. NOTE: Testing is not required unless mandated by the local health authority. Participants with HIV infection may be eligible if ALL of the following are applicable:

   1. Receiving an approved, stable, effective combination antiretroviral therapy regimen for > 3 months prior to the planned first study intervention. NOTE: please review Section 5.7 and consider whether any actions should be taken to minimize potential drug-drug interactions,
   2. CD4 T cell count > 350 cells/µl,
   3. CD4 T cell nadir (lowest historical count) > 200 cells/µl, and
   4. Viral load confirmed as < 50 copies/mL during Screening.
9. Participants with a known history of chronic viral infections as indicated below. NOTE: Testing for hepatitis B virus (HBV) or hepatitis C virus (HCV) is not required unless mandated by the local health authority.

   1. Known HBV infection defined as hepatitis B surface antigen reactive. NOTE: Participants with HBV infection on stable anti-viral therapy for > 4 weeks prior to the planned first study intervention and viral load confirmed as undetectable during Screening may be eligible.
   2. Known active HCV infection defined as detectable HCV RNA (qualitative) infection. NOTE: History of HCV is not exclusionary if participants have received curative treatment and viral load is confirmed as undetectable during screening.
10. Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type.
11. Any medical condition that would, in the investigator's or Sponsor's judgement, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Regression of primary uveal melanoma after Tebentafusp treatment in 20% of treated patients. | 3 months post-eye treatment
  Regression is defined as ≥ 20% reduction in tumor volume. All estimates of rates will be presented with corresponding 95% exact confidence intervals. For regression rate, the method of Atkinson and Brown will be used to allow for the two-stage design.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 5 years
  Will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events (AE) version 5.0. All estimates of rates will be presented with corresponding 95% exact confidence intervals. AEs will be reported for each dose level and presented as tables of frequency of AEs by body system and by worse severity grade observed. AE term start and end date, severity, seriousness, outcome, action taken regarding study drugs and relationship to each study drug will also be reported. The summary tables will also discuss AEs leading to death and AEs leading to study drug(s) discontinuation. Tables should indicate related and unrelated events. Laboratory data will be presented by dose level at each observation time. Values outside normal limits will be identified and summarized by frequency distribution.
Detection of plasma circulating tumor-derived deoxyribonucleic acid (ctDNA) and correlation of antitumor response | 22 months
  Plasma of patients will be collected for all patients at baseline (within 28 days of first dose), cycle 2 day 1, post-tebentafusp (within 14 days of last dose), and at the 3 month post-treatment evaluation. ctDNA response will be measured (defined as ≥0.3 log reduction) in ctDNA-evaluable patients as measured using Signatera assay and correlated with eye tumor regression.
Detection of aqueous humor ctDNA and correlation of antitumor response | 22 months
  Aqueous humor of patients will be collected at baseline and post-tebentafusp; if no ctDNA is detectable in the aqueous humor after 5 patients we will stop collecting aqueous ctDNA for the rest of the patients. ctDNA response will be measured (defined as ≥0.3 log reduction) in ctDNA-evaluable patients as measured using Signatera assay and correlated with eye tumor regression.

OTHER OUTCOMES:
Assessment of visual acuity loss at baseline (prior to Tebentafusp treatment), prior to plaque brachytherapy, and 3) following plaque brachytherapy (after resolution of any radiation side effects/edema). | 22 months
  Ophthalmological examination for assessment of disease: this will be performed within 48 hours prior to Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 2 Day 1. Additional ophthalmological examinations may be performed if clinically indicated. All ophthalmological examinations must be performed and interpreted by a qualified ocular oncologist. Examination will include clinical eye examination, ophthalmic ultrasound, wide-angle fundus imaging, and optical coherence tomography
Change in radiation dose to the fovea. | 22 months
  Change in modeled radiation dose at critical eye structures before and after neoadjuvant Tebentafusp therapy
Enucleation vs plaque brachytherapy post-treatment | 22 months
  Assessment of proportion of patients who had planned enucleation prior to therapy, but following Tebentafusp treatment were suitable for plaque brachytherapy.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No